CLINICAL TRIAL: NCT03053375
Title: The Effect of Pulsed Electromagnetic Field Therapy on Patients With Low Back Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Bridgeport (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2015-05-03
Record Dates: First submitted 2017-02-06; First posted 2017-02-15 (Actual); Last update posted 2017-02-15 (Actual); Status verified 2017-02

CONDITIONS: Low Back Pain
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (4):
- Acute/subacute; active device (Experimental): MDCure active device
  Interventions: Device: MDCure
- Acute/subacute; sham (Placebo Comparator): MDCure sham device
  Interventions: Device: MDCure
- Chronic; active device (Experimental): MDCure active device
  Interventions: Device: MDCure
- Chronic; sham (Placebo Comparator): MDCure sham device
  Interventions: Device: MDCure

INTERVENTIONS:
Device: MDCure — Battery powered portable pulsed electromagnetic therapy device

SUMMARY:
This study will examine the effects of a portable of pulsed electromagnetic field (PEMF) device (MD Cure, Aerotel, USA) compared with a sham device on patient-reported outcomes of pain and function in patients with either acute/subacute or chronic low back pain (LBP).

DETAILED DESCRIPTION:
This study is a double-blind, placebo-controlled, randomized pilot study comparing usual care + PEMF with usual care + sham.

The investigators will recruit patients with LBP from the University of Bridgeport chiropractic clinic, and will enroll 80 total subjects: 40 with acute or subacute LBP, and 40 with chronic LBP. Within each of those populations the investigators will assign 20 subjects to receive usual care + PEMF, and 20 to receive usual care + sham. The investigators will track any other treatments initiated or discontinued during the trial.

Patients who agree to participate with be randomly given a functional PEMF device or a sham unit. Patients and clinicians will be blinded to the assignment. All subjects will be given the same instructions for daily use of the devices, and will continue to receive usual follow-up at the UBCC clinic as indicated. The investigators will collect patient-reported measures of pain and function pain at baseline, 6 weeks, and 12 weeks, and will collect data on adverse effects at each visit and at 6 and 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* UBCC patient
* complaint of LBP intensity 4/10 or greater on the Numerical Rating Scale
* diagnosis of a mechanical LBP condition
* age 18-70 years
* fluency in written and spoken English
* for female subjects, be postmenopausal, surgically sterile, abstinent, or agree to practice an effective method of birth control for the duration of the study if sexually active
* a willingness to participate in the study as evidenced by a signed informed consent form

Exclusion Criteria:

* current LBP complaint of 3/10 or less on the Numerical Rating Scale
* diagnosis or suspicion of LBP caused by cancer, infection, referred visceral pain, inflammatory arthropathy, or other non-mechanical process
* current or planned pregnancy
* any electrically-based implanted devices such as pacemakers defibrillators, spinal cord stimulators, insulin pumps; metallic implants (e.g. surgical fusion constructs, disc replacements) in the low back
* status post any lumbosacral spine surgery; significant mental health co-morbidities such as severe depression, schizoaffective disorders, suicidal ideation
* inability to understand and/or complete all components of the informed consent process without the assistance of another person (e.g. without proxy)
* inability to adhere to and comply with the treatment protocol.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-02-08 (Actual); Primary Completion 2017-08-30 (Estimated); Study Completion 2018-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in pain intensity | Baseline, weeks 6 and 12
  Numerical Rating Scale
Change in low back pain related disability | Baseline, weeks 6 and 12
  Oswestry Disability Index

CONTACTS AND LOCATIONS:
Locations (1):
- University of Bridgeport, Bridgeport, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Lisi AJ, Scheinowitz M, Saporito R, Onorato A. A Pulsed Electromagnetic Field Therapy Device for Non-Specific Low Back Pain: A Pilot Randomized Controlled Trial. Pain Ther. 2019 Jun;8(1):133-140. doi: 10.1007/s40122-019-0119-z. Epub 2019 Mar 12. PMID 30868475